CLINICAL TRIAL: NCT00814918
Title: Topical 5-ALA-PDT With Blu-U Therapy Vs. Topical 5-ALA With Pulse Dye Laser In Treatine Recalcitrant Acne Vulgaris
Brief Title: Topical 5-ALA-PDT With Blu-U Therapy Versus Topical 5-ALA With Pulse Dye Laser In Treating Recalcitrant Acne Vulgaris
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15929B
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; acne; dermatalogy
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 5-ALA Application and exposure using Blu-U light to 1/2 of face.
  Interventions: Drug: 5-ALA with Blu-U Light
- 2 (Experimental): 5-ALA Application and exposure using Candela V-beam Pulse Dye Laser to 1/2 of face.
  Interventions: Drug: 5-ALA with Candela V-beam Pulse Dye Laser

INTERVENTIONS:
Drug: 5-ALA with Blu-U Light — 20% 5-ALA Levulan Kerastick will be crushed and prepared for application after shaking for at least 3 minutes. Topical 5-ALA will be applied liberally on skin with extra pressure on lesions.Skin will be exposed to DUSA Blu-U light (417nm).
  Arms: 1
Drug: 5-ALA with Candela V-beam Pulse Dye Laser — 20% 5-ALA Levulan Kerastick will be crushed and prepared for application after shaking for at least 3 minutes. Topical 5-ALA will be applied liberally on skin with extra pressure on lesions.Skin will be exposed to Candela V-beam Pulsed Dye Laser (595 nm).
  Arms: 2

SUMMARY:
The goal of this study is to compare how efficient two different types of PDTs are when used in combination with topical 5-ALA. The two types of PDT lights are Blu-U light and Candela V-beam Pulse Dye Laser.

ELIGIBILITY:
Inclusion Criteria:

* 18-79 years of age
* Patients who failed the topical and oral antibiotics after 6 month therapy.
* Patients who failed the topical retinoids after 6 month therapy.
* Patients that are not good candidate to start oral isotretinoin (Accutane) due to contraindications.

Exclusion Criteria:

* Patients who have had Isotretinoin therapy less that 1 year prior to this ALA-PDT procedure.
* Patients who have an adverse reaction to light exposure (for example photo- exacerbated seizures).
* Patients with a history of porphyria.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Acne complete /incomplete therapy and reoccurence | 18 months

SECONDARY OUTCOMES:
Early skin responses 2 weeks post therapy (erythema, scaling, post inflammatory skin changes, fine wrinkling of skin, mottled pigmentation) | 2-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Tsoukas, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States